CLINICAL TRIAL: NCT06682611
Title: An, Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of SYHA1813 Single Agent or in Combination With Different Regimens in Unresectable Locally Advanced or Metastatic Solid Tumors.
Brief Title: Safety and Efficacy of SYHA1813 Single Agent or in Combination With Different Regimens in Unresectable Locally Advanced or Metastatic Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1814-005
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Unresectable Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Carboplatin; Cisplatin; Paclitaxel; Etoposide; Everolimus; regorafenib

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-center, multi-cohort, phase Ib/II clinical trial, divided into 8 cohorts according to tumor types. Cohorts 1-4 are SYHA1813 combined with different regimens, including safety run-in stage and cohort expansion stage. Cohorts 5-8 are SYHA1813 monotherapy and only include the expansion cohorts. In the expansion stage, cohorts 1-6 are single-arm studies, cohorts 7-8 are randomized controlled studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYHA1813 single agent or in combination with different regimens (Experimental): Cohorts 1-4 are SYHA1813 combined with different regimens. Cohorts 5-8 are SYHA1813 monotherapy.
  Interventions: Drug: SYHA1813; Drug: Everolimus; Drug: Regorafenib
- Control group (Active Comparator): The cohort 7 control group is Everolimus. The cohort 8 control group is Regorafenib.
  Interventions: Drug: SYHA1813; Drug: SG001; Drug: HB1801; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Etoposide; Drug: Everolimus; Drug: Regorafenib

INTERVENTIONS:
Drug: SYHA1813 — In accordance with the protocol
Drug: SG001 — In accordance with the protocol
  Arms: Control group
Drug: HB1801 — In accordance with the protocol
  Arms: Control group
Drug: Carboplatin — In accordance with the protocol
  Arms: Control group
Drug: Cisplatin — In accordance with the protocol
  Arms: Control group
Drug: Paclitaxel — In accordance with the protocol
  Arms: Control group
Drug: Etoposide — In accordance with the protocol
  Arms: Control group
Drug: Everolimus — In accordance with the protocol
Drug: Regorafenib — In accordance with the protocol

SUMMARY:
This is an open-label, multi-center, multi-cohort, phase Ib/II clinical trial, divided into 8 cohorts according to tumor types. Cohorts 1-4 are SYHA1813 combined with different regimens, including safety run-in stage and cohort expansion stage. Cohorts 5-8 are SYHA1813 monotherapy and only include the expansion cohorts. The primary objective was to evaluate the safety and efficacy of SYHA1813 single agent or in combination with different regimens in unresectable locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
In the safety run-in stage, the "3+3" design is used to evaluate the tolerability and safety of different dose levels combined with different regimens, and the observation period of DLT is set as the first treatment cycle. After 3 DLT-evaluable participants at each dose level completed the DLT observation period, the safety of the dose level is evaluated by an SMC consisting of the investigator and the sponsor's medical monitor. Cohorts 1-4 enter the cohort expansion stage after determining the SYHA1813 dose regimen during the safety run-in stage. Cohorts 5-8 enter the cohort expansion stage directly. In the expansion stage, cohorts 1-6 are single-arm studies, the primary endpoint is ORR as evaluated by investigator according to RECIST 1.1. Cohorts 7-8 are randomized controlled studies, the primary endpoint is PFS as evaluated by investigator according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >= 18 years;
2. Unresectable locally advanced or metastatic solid tumors confirmed by histology or cytology:
3. There is at least one measurable lesion in the baseline period (RECIST1.1);
4. ECOG PS of 0-1;
5. The expected survival time is >=3 months;
6. The organ function level and related laboratory indicators must meet the following requirements (No blood transfusion or hematopoietic stimulating factor therapy received within 14 days prior to the first medication (queue 1 to 6)/prior to randomization (queue 7 and queue 8):

   ANC≥1.5×10^9/L； PLT≥100×10^9/L（Liver cancer patients PLT≥75×10^9/L）； Hb≥90 g/L； TBIL≤1.5×ULN，and for Gilbert's syndrome, liver cancer or liver metastasis patients TBIL≤3×ULN； ALT和AST≤2.5×ULN，for liver cancer or liver metastasis patients ≤5×ULN； Child-Pugh Grade A (only applicable to queue 8)； ALB≥30 g/L； Cr≤1.5×ULN，IF Cr>1.5×ULN，Ccr≥60 mL/min（Cockcroft-Gault）is required； APTT and INR≤1.5×ULN
7. The subjects must agree to take medically approved contraceptive measures for at least 6 months from the beginning of the study to the last dose of drug.

Exclusion Criteria:

1. Patients who are known or suspected to be allergic to the test drug or its components;
2. Excluding the disease studied in this trial, there are other primary malignant tumors that have progressed or require treatment within the past 3 years prior to screening (except for effectively controlled skin basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer or cured breast carcinoma in situ);
3. The toxicity of previous anti-tumor treatments has not recovered (≤grode 1), except for hair loss and other adverse reactions judged by the investigator that do not affect the safety of the study medication;
4. Active leptomeningeal disease or CNS metastases that are not well controlled;
5. Uncontrollable active infections occurred within 14 days prior to the first medication (queue 1 to 6)/prior to randomization (queue 7 and queue 8), requiring systemic treatment with intravenous antibiotic infusion
6. Patients with evidence of bleeding tendency or medical history within 28 days;
7. Patients have risk factors for intestinal obstruction or intestinal perforation;
8. The subject has poorly healed wounds, ulcers or fractures;
9. Urine protein ≥ 2+, and 24-hour urine protein quantitative ≥ 1.0g/24h;
10. Patients have large pleural effusions, pericardial effusions, or abdominopelvic effusions;
11. Human immunodeficiency virus (HIV) antibody positive; active hepatitis C, with antibody positive and HCV RNA test positive; active hepatitis B, with HBsAg positive, and HBV-DNA value>500 IU/ml or 2500 copies/mL;
12. Has a history of active tuberculosis;
13. History of interstitial lung disease (except for radiotherapy-induced focal interstitial pneumonia), noninfectious pneumonitis requiring glucocorticoid therapy;
14. Received immunosuppressants such as PD-1 or PD-L1 inhibitors in the recurrent or metastatic phase (only for Cohort 1);
15. Prior treatment with a VEGFR-TKI inhibitor or other anti-angiogenic agent (except for Cohort 5,7,8);
16. Pregnant or lactating women;
17. Participants who may have poor compliance as judged by the investigator, such as a clear history of neurological or psychiatric disorders (including epilepsy or dementia), current psychiatric disorders, psychotropic drug abuse, etc.;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-11-13 (Estimated); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-11-13 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to approximately 2years
  Safety run-in stage，Dose-limiting toxicity (DLT) will be assessed according to NCI-CTCAE v5.0.
Frequency and severity of TEAE and SAE | Up to approximately 2years
  Safety run-in stage
ORR | Up to approximately 2 years
  Cohorts 1-6, Objective response rate (ORR) as evaluated by Investigator (RECIST1.1)
PFS | Up to approximately 2years
  Cohorts 7-8, Progression-free survival (PFS) as evaluated by Investigator (RECIST1.1)

SECONDARY OUTCOMES:
OS | Up to approximately 2years
  Overall survival
DoR | Up to approximately 2years
  Duration of response
DCR | Up to approximately 2 years
  Disease control rate
Frequency and severity of TEAE and SAE | Up to approximately 2 years
  Safety
Plasma Concentration | Up to approximately 2 years
  Concentration of SYHA1813/SG001/HB1801 in serum
Immunogenicity | Up to approximately 2 years
  Incidence of SG001 Anti-drug antibody (ADA) and neutralizing antibody (Nab) (if applicable)

IPD SHARING:
Plan to Share IPD: No